CLINICAL TRIAL: NCT03923855
Title: Clinical Evaluation of the BTL-899 Device for Non-invasive Lipolysis on Human Fat Tissue
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: BTL Industries Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 899-H1
Record Dates: First submitted 2019-04-18; First posted 2019-04-23 (Actual); Last update posted 2019-12-20 (Actual); Status verified 2019-12

CONDITIONS: Improvement of Abdomen Appearance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BTL-899 Therapy Arm (Experimental)
  Interventions: Device: BTL-899

INTERVENTIONS:
Device: BTL-899 — BTL-899 therapy

SUMMARY:
The subjects will be enrolled and assigned to a single study group. They will be required to complete two treatment visits and come for a biopsy procedure.

ELIGIBILITY:
Inclusion Criteria:

* Age above 21 years and below 60 years
* Voluntarily signing of the informed consent form
* Women of child-bearing potential are required to use birth control measures during the whole duration of the study
* Eligibility to fat tissue biopsy at surgeon discretion, incl. at least 3-4 cm pinchable fat in the abdominal area
* Subjects willing and able to abstain from partaking in any procedure to promote body contouring during study participation
* Subjects willing and able to maintain his/her regular (pre-procedure) diet and exercise regimen without effecting significant change in either direction during study participation

Exclusion Criteria:

* Electronic implants (such as cardiac pacemakers, defibrillators and neurostimulators)
* Cardiovascular diseases
* Disturbance of temperature or pain perception
* Pulmonary insufficiency
* Metal implants
* Drug pumps
* Malignant tumor
* Hemorrhagic conditions
* Septic conditions and empyema
* Acute inflammations
* Systemic or local infection such as osteomyelitis and tuberculosis
* Contagious skin disease
* Elevated body temperature
* Pregnancy
* Breastfeeding
* Injured or otherwise impaired muscles
* Scars, open lesions and wounds at the treatment area
* Basedow's disease
* Previous liposuction in the treatment area in the last six months
* Abdominal wall diastasis
* Unstable weight within the last 6 months (change in weight ± 3%)
* Previous body contouring treatments in the abdomen area in the last three months
* Any disease or condition contradicting the fat tissue biopsy at the surgeon discretion
* Any disease or condition that may compromise the histologic observation at the pathologist discretion

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2019-09-17 (Actual); Study Completion 2019-10-07 (Actual)

PRIMARY OUTCOMES:
Histology Examination | 4 months
  Histological examination of the fat tissue after BTL-899 treatment at various days after the procedure
Evaluation of Satefy: Occurence of adverse events throughout the study | 4 months
  Following the occurence of adverse events throughout the study.

CONTACTS AND LOCATIONS:
Locations (1):
- Dr. Denkova Dermatology, Sofia, Bulgaria